CLINICAL TRIAL: NCT03312244
Title: Study of the Role of Peripheral Acetylcholinesterase Inhibitor Pyridostigmine as Immunomodulators in a Population of Patients Living With Human Immunodeficiency Virus Infection.
Brief Title: Pyridostigmine as Immunomodulator in People Living With HIV
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to COVID-19, effective 3/19/2020 recruitment is halted until further notice
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Sergio I. Valdés-Ferrer, MD, PhD, Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ref. 1873
Record Dates: First submitted 2017-04-01; First posted 2017-10-17 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: HIV-1-infection; CD4+ T Lymphocytopenia; Immune Deficiency; Immuno-senescence
MeSH Terms: conditions — T-Lymphocytopenia, Idiopathic CD4-Positive; Immunologic Deficiency Syndromes | interventions — Pyridostigmine Bromide; Starch

STUDY DESIGN:
Intervention Model Description: 12x12 weeks of pyridostigmine or placebo followed by crossing-over to the other arm of intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants will be blinded. The steering committee will have the authority to open the blinding in case of adverse effects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pyridostigmine (Experimental): Pyridostigmine 180mg/d slow-release formulation
  Interventions: Drug: Pyridostigmine Bromide
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyridostigmine Bromide — Pyridostigmine 180mg/day p.o.
  Other Names: Mestinon Timespan
  Arms: Pyridostigmine
Drug: Placebo — Placebo
  Other Names: Starch (pharmaceutical grade)
  Arms: Placebo

SUMMARY:
Human immunodeficiency virus (HIV) infection is characterized by persistent immune activation and a constant turnover of T cells. This leads to a precipitous fall in the number of T cells, as well as to an early immunosenescence. This results in increased susceptibility to opportunistic infections. In these patients, modulation of the immune response represents a promising mechanism to maintain immunological homeostasis and prevent the development of pathology. We hypothesize that the addition of pyridostigmine to the regular combined antiretroviral therapy will result in a decrease in T cell overactivation and a reduction in circulating inflammatory markers.

DETAILED DESCRIPTION:
Human immunodeficiency virus (HIV) infection is a public health problem with enormous personal, and social losses. According to the National Mexican HIV/AIDS survey, more than 235,000 new cases of HIV infection were reported in Mexico between 1983 and 2015.

HIV infection is characterized by persistent immune activation and a constant turnover of T cells. This leads to a precipitous fall in the number of CD4+ and CD8+ T cells, as well as to early immunosenescence. This immunosenescence results in increased susceptibility to opportunistic infections and a profound decrease in circulating and mucosal T cells. In these patients, modulation of the immune response represents a promising mechanism to maintain immunological homeostasis and prevent the development of pathology. From this perspective, it is posible that a reduced immune activation -rather than accelerating the progression of infection- may be an important factor in controlling infection and delaying the progression from chronic infection to acquired immunodeficiency syndrome (AIDS).

The administration of combined antiretroviral therapy (cART) has resulted in a reduction in the mortality of these patients, although the occurrence of late morbidity due to both infection and treatment has increased. Unfortunately, even in countries with complete coverage for HIV-infection, a large group of patients do not start treatment until late stages, in which immunosenescence is profound and the possibilities of immunological recovery (increase in T cell counts CD4+, normalization of the CD4+/CD8+ index, decrease in susceptibility to opportunists, normalization in the cellular response to vaccines) are very low. In this context, finding new immuno-modulatory strategies that are both easily applicable and potentially improving survival and quality of life is crucial.

The therapeutic use of neuroimmune regulators in HIV infection has been poorly explored. The nervous system has evolutionary mechanisms of reflex control of the inflammatory response, such as cholinergic anti-inflammatory pathway. Cholinergic stimulation through the use of nicotinic agonists has shown promising effects in murine and cellular models of systemic inflammation. Since cholinergic agonists are rapidly degraded or cause side effects, we performed a pilot study using pyridostigmine (Mestinon®), an acetylcholinesterase inhibitor (ACh-E), in HIV-infected patients. We observed that administration of pyridostigmine decreases the activation and proliferation of HIV-infected T cells, reduces the production of interferon (IFN)-γ and increases that of interleukin (IL)-10 (Valdés-Ferrer SI et al., AIDS Research And Human Retrovir 2009). In a second open-label pilot study in seven chronically infected patients with full virologic suppression but without concomitant elevation of CD4+ T cell counts, we found that the addition of pyridostigmine to ART led to a sustained and significant increase in the number of CD4 + T cells (PRS record: NCT00518154; Valdés-Ferrer SI, et al., Frontiers in Immunology, 2017). These results suggest that the addition of pyridostigmine to antiretroviral therapy may be beneficial in achieving and maintaining immunological homeostasis in patients with HIV.

The present study will address the potential effectiveness of add-on pyridostigmine (180mg, once per day, P.O.) on CD4+ T cell counts, CD4+/CD8+ ratio, as well as ex-vivo markers of T cell phenotype and activity. The study is designed as a 24-week crossover study where patients will start a 12-week of pyridostigmine or placebo, and then crossing-over for an additional 12 weeks (placebo-to-pyridostigmine, and pyridostigmine-to-placebo).

Since pyridostigmine is a commonly used drug for both myasthenia gravis and as a preventive in biological warfare cases, if our hypotheses are correct, the results can be easily extrapolated to clinical practice, as there is enough long-term evidence of utility and safety of the drug.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected subjects 18 years of age or older
2. Receiving stable ART for at least six months
3. At least two undetectable viral load determinations in the previous six months
4. Patient agrees to participate and signs informed consent

Exclusion Criteria:

1. Concomitant active infectious or neoplastic disease
2. History of new AIDS-defining events in the previous six months
3. If a participant is female, pregnancy or breast-feeding
4. Exposure to an investigational agent, chemotherapy or radiotherapy within the previous 28 days
5. Currently taking or planning to take treatment for Tuberculosis
6. Being unable to follow or comply with the protocol interventions
7. The participant is receiving immunosuppressive treatment, including corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
CD4+ T cell count | Change from baseline, at 12 and 24 weeks
  Change in total CD4+ T cel count from baseline

SECONDARY OUTCOMES:
soluble CD14 receptor | Change from baseline, at 12 and 24 weeks
  Change in circulating (plasma) soluble CD14 receptor from baseline
CD4+ / CD8+ | Change from baseline, at 12 and 24 weeks
  Change in index of CD4+ to CD8+ T cells from baseline
Inteleukin (IL)-6 | Change from baseline, at 12 and 24 weeks
  Change in circulating (plasmatic) IL-6 from baseline
TREC levels | Change from baseline, at 12 and 24 weeks
  Changes in T cell receptor excision DNA circle (TREC) levels

CONTACTS AND LOCATIONS:
Overall Officials: Juan Sierra-Madero, MD, Study Director — INNSZ
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: Yes
All data will be freely available to all research parties involved
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available after finishing with recruitment.
Access Criteria: Data will be made available by request.

REFERENCES:
- [Result] Autran B, Carcelain G, Li TS, Blanc C, Mathez D, Tubiana R, Katlama C, Debre P, Leibowitch J. Positive effects of combined antiretroviral therapy on CD4+ T cell homeostasis and function in advanced HIV disease. Science. 1997 Jul 4;277(5322):112-6. doi: 10.1126/science.277.5322.112. PMID 9204894
- [Result] Pakker NG, Notermans DW, de Boer RJ, Roos MT, de Wolf F, Hill A, Leonard JM, Danner SA, Miedema F, Schellekens PT. Biphasic kinetics of peripheral blood T cells after triple combination therapy in HIV-1 infection: a composite of redistribution and proliferation. Nat Med. 1998 Feb;4(2):208-14. doi: 10.1038/nm0298-208. PMID 9461195
- [Result] Kaufmann GR, Perrin L, Pantaleo G, Opravil M, Furrer H, Telenti A, Hirschel B, Ledergerber B, Vernazza P, Bernasconi E, Rickenbach M, Egger M, Battegay M; Swiss HIV Cohort Study Group. CD4 T-lymphocyte recovery in individuals with advanced HIV-1 infection receiving potent antiretroviral therapy for 4 years: the Swiss HIV Cohort Study. Arch Intern Med. 2003 Oct 13;163(18):2187-95. doi: 10.1001/archinte.163.18.2187. PMID 14557216
- [Result] Corbeau P, Reynes J. Immune reconstitution under antiretroviral therapy: the new challenge in HIV-1 infection. Blood. 2011 May 26;117(21):5582-90. doi: 10.1182/blood-2010-12-322453. Epub 2011 Mar 14. PMID 21403129
- [Result] Moore DM, Hogg RS, Yip B, Wood E, Tyndall M, Braitstein P, Montaner JS. Discordant immunologic and virologic responses to highly active antiretroviral therapy are associated with increased mortality and poor adherence to therapy. J Acquir Immune Defic Syndr. 2005 Nov 1;40(3):288-93. doi: 10.1097/01.qai.0000182847.38098.d1. PMID 16249702
- [Result] Piconi S, Trabattoni D, Gori A, Parisotto S, Magni C, Meraviglia P, Bandera A, Capetti A, Rizzardini G, Clerici M. Immune activation, apoptosis, and Treg activity are associated with persistently reduced CD4+ T-cell counts during antiretroviral therapy. AIDS. 2010 Aug 24;24(13):1991-2000. doi: 10.1097/QAD.0b013e32833c93ce. PMID 20651586
- [Result] Tracey KJ. Physiology and immunology of the cholinergic antiinflammatory pathway. J Clin Invest. 2007 Feb;117(2):289-96. doi: 10.1172/JCI30555. PMID 17273548
- [Result] Valdes-Ferrer SI, Crispin JC, Belaunzaran PF, Cantu-Brito CG, Sierra-Madero J, Alcocer-Varela J. Acetylcholine-esterase inhibitor pyridostigmine decreases T cell overactivation in patients infected by HIV. AIDS Res Hum Retroviruses. 2009 Aug;25(8):749-55. doi: 10.1089/aid.2008.0257. PMID 19645607
- [Result] Ku NS, Song YG, Han SH, Kim SB, Kim HW, Jeong SJ, Kim CO, Kim JM, Choi JY. Short communication: factors influencing time to CD4(+) T cell counts >200 cells/mm(3) in HIV-infected individuals with CD4(+) T cell <50 cells/mm(3) at the time of starting combination antiretroviral therapy. AIDS Res Hum Retroviruses. 2012 Dec;28(12):1594-7. doi: 10.1089/AID.2011.0282. Epub 2012 Jun 25. PMID 22632127
- [Result] Kawashima K, Fujii T. The lymphocytic cholinergic system and its biological function. Life Sci. 2003 Mar 28;72(18-19):2101-9. doi: 10.1016/s0024-3205(03)00068-7. PMID 12628464
- [Result] Rosas-Ballina M, Olofsson PS, Ochani M, Valdes-Ferrer SI, Levine YA, Reardon C, Tusche MW, Pavlov VA, Andersson U, Chavan S, Mak TW, Tracey KJ. Acetylcholine-synthesizing T cells relay neural signals in a vagus nerve circuit. Science. 2011 Oct 7;334(6052):98-101. doi: 10.1126/science.1209985. Epub 2011 Sep 15. PMID 21921156
- [Result] Valdes-Ferrer SI, Crispin JC, Belaunzaran-Zamudio PF, Rodriguez-Osorio CA, Cacho-Diaz B, Alcocer-Varela J, Cantu-Brito C, Sierra-Madero J. Add-on Pyridostigmine Enhances CD4+ T-Cell Recovery in HIV-1-Infected Immunological Non-Responders: A Proof-of-Concept Study. Front Immunol. 2017 Oct 18;8:1301. doi: 10.3389/fimmu.2017.01301. eCollection 2017. PMID 29093707